CLINICAL TRIAL: NCT03773367
Title: Irinotecan-based Triplet (FOLFOXIRI) as Perioperative Treatment in Resectable Gastric and Gastroesophageal Junction Adenocarcinoma.
Acronym: INTENSE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEGCG18-01
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Resectable Gastric and Gastroesophageal Junction Adenocarcinoma
Keywords: Gastric adenocarcinoma; Gastroesophageal junction adenocarcinoma; Chemotherapy; Fluorouracil; Oxaliplatin; Irinotecan; Preoperative chemotherapy; Postoperative chemotherapy; Histopathological response; Rate of R0-resection
MeSH Terms: interventions — Fluorouracil; Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with chemotherapy pre- and postoperative. (Experimental)
  Interventions: Drug: Fluorouracil; Drug: Oxaliplatin; Drug: Irinotecan

INTERVENTIONS:
Drug: Fluorouracil — Treatment with Fluorouracil, Oxaliplatin, and Irinotecan is given for 4 cycles pre- and postoperatively, in total 8 cycles.
Drug: Oxaliplatin — Treatment with Fluorouracil, Oxaliplatin, and Irinotecan is given for 4 cycles pre- and postoperatively, in total 8 cycles.
Drug: Irinotecan — Treatment with Fluorouracil, Oxaliplatin, and Irinotecan is given for 4 cycles pre- and postoperatively, in total 8 cycles.

SUMMARY:
In this clinical trial, patients with gastric and gastroesophageal junction adenocarcinoma will be included. Treatment with curative intent will be given with chemotherapy for 4 cycles with fluorouracil, oxaliplatin and irinotecan preoperatively followed by surgery, and then additionally 4 cycles of the same chemotherapy postoperatively. The standard treatment today is preoperative treatment with fluorouracil and oxaliplatin pre-and postoperatively. The rationale for this trial is, that the addition of irinotecan might improve treatments results.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified, resectable gastric or gastroesophageal (GE) (gastroesophageal) junction (Siewert type I-III) adenocarcinoma Confirmation of patient operability by surgeon
* Primary tumor, regional nodes, metastasis (TNM), 8th edition): cT2-4a or cN+, cM0
* Age: 18 years or older
* World Health Organization (WHO) performance status ≤ 1
* Exclusion of peritoneal carcinomatosis (if clinically suspected) via laparoscopy
* Adequate laboratory findings:

  * hematological: hemoglobin > 90 g/L (transfusion is allowed to attain this), absolute neutrophil count (ANC) ≥ 1,5 x 109/L, platelets ≥ 75 x 109/L
  * hepatic: bilirubin ≤ 1.5 x upper limit of normal (ULN), alanine aminotransferase (ALAT) ≤ 3 x ULN
  * renal: creatinine ≤ 1.5 x ULN (upper limit of normal)
* Fertile men and women must use highly effective means of contraception (failure rate <1%) such as:

  * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal administration)
  * progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable administration)
  * intrauterine device
  * intrauterine hormone-releasing system
  * bilateral tubal occlusion
  * vasectomised partner
  * sexual abstinence
* Signed written informed consent
* The patient must be able to comply with the protocol

Exclusion Criteria:

* Neuroendocrine or adenosquamous carcinoma
* Prior oncological treatment or surgical resection for the present disease
* Presence of other concurrent malignancies or previous malignancies within 5 years except for adequately treated basal or squamous cell carcinoma of the skin or in-situ carcinoma of the cervix uteri
* Clinically significant (i.e. active) cardiovascular disease e.g. myocardial infarction (≤ 6 months), unstable angina, New York Heart Association (NYHA) grade III-IV congestive heart failure
* Active inflammatory bowel disease
* Symptomatic peripheral neuropathy greater than grade 1 (CTCAE version 4.03)
* Known hypersensitivity to any contents of the study drugs
* Pregnancy (positive pregnancy test) and/or breast feeding
* Any other serious or uncontrolled illness which in the opinion of the investigator makes it undesirable for the patient to enter the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-12-14 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
To determine the rate of histopathological response according to Becker criteria. | After surgery.
  Assessment of histopathological response, ypTNM, resection margin and residual tumor status. If Laurén classification and mismatch repair (MMR) or microsatelite instability status (MSI) could not be assessed on pretreatment biopsies it should be assessed on the resected specimen. Results do not have to be awaited before start of chemotherapy.

CONTACTS AND LOCATIONS:
Locations (4):
- Oslo University Hospital, Ullevål Hospital, Oslo, Norway
- Sweden (3):
  - Lund University Hospital, Lund
  - Karolinska University Hospital, Stockholm
  - Centrallasarettet i Växjö, Vaxjo

IPD SHARING:
Plan to Share IPD: No